CLINICAL TRIAL: NCT00821262
Title: Sevoflurane and Cardiac Protection in High Risk Patients Undergoing Cardiac Surgery. A Randomized Controlled Study.
Brief Title: Sevoflurane in Cardiac Surgery
Acronym: SEVO AIFA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Giovanni Landoni, DM, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GO/URC/ER/mm 412/DG
Record Dates: First submitted 2009-01-12; First posted 2009-01-13 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Anesthesia; Cardiac Surgery
Keywords: Sevoflurane; Anesthesia; Troponin; Myocardial Preconditioning; Surgery, Cardiac; Stents; Non-cardiac Surgery; Surgery
MeSH Terms: interventions — Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- sevoflurane (Experimental): The study group will receive Sevoflurane for a 4-6 hours period (from anesthesia induction to transfer to ICU).
  Interventions: Drug: sevoflurane
- propofol (Active Comparator): The control group will receive propofol for the same 4-6 hours period.
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: sevoflurane
  Arms: sevoflurane
Drug: propofol
  Arms: propofol

SUMMARY:
Patients undergoing high risk cardiac surgery (combined CABG and valvular procedures) will be randomized to receive a total intravenous anesthesia or an anesthesia plan with sevoflurane.

The investigators want to document whether the cardioprotective properties of volatile agents could translate in an improved outcome after cardiac surgery in high risk patients.

DETAILED DESCRIPTION:
Background

It is commonly believed that the choice of the primary anesthetic agent does not result in different outcomes after cardiac surgery. Recent evidence however has indicated that volatile anesthetics improve post-ischemic recovery. These results have been summarized in a meta-analysis of 22 randomized studies, involving 1922 patients: the use of volatile anesthetics was associated with significant reductions of myocardial infarctions (24/979 [2.4%] in the volatile anesthetics group vs 45/874 [5.1%] in the control arm, odds ratio [OR]=0.51 [0.32-0.84], and mortality (4/977 [0.4%] vs 14/872 [1.6%], OR=0.31 [0.12-0.80].

Furthermore, the use of volatile anesthetics was associated with shorter intensive-care unit stay (WMD=-7.10 hours [-11.47; -2.73], and time to hospital discharge (WMD=-2.26 days [-3.83; -0.68].

All the studies of the meta-analysis included low risk patients undergoing isolated procedures (mostly coronary artery bypass grafting).

Objectives

Investigators are planning a large multicentre randomized controlled study to confirm the beneficial cardioprotective effects of volatile anesthetics in cardiac surgery as indicated by a reduced intensive care stay and/or death in an high risk population of patients undergoing combined valvular and coronary procedures. Secondary endpoints will be: cardiac troponin release; incidence of myocardial infarction; time on mechanical ventilation; postoperative hospital stay

Methods

Various centers will randomize 200 patients to receive either a total intravenous anesthesia with propofol or an anesthesia with sevoflurane. All patients will receive a standard middle dose opiates anesthesia. All the perioperative management will be otherwise identical and standardized. Transfer out of the intensive care will be performed with SpO2 94% or greater at an FiO2 of 0.5 or less by facemask, adequate cardiac stability with no hemodynamically significant arrhythmias, chest tube drainage less than 50 ml/h, urine output greater than 0.5 ml/kg/h, no intravenous inotropic or vasopressor therapy in excess of dopamine 5 ug/kg/min, and no seizure activity.

Expected Results

The reduced cardiac damage (reduction in cardiac troponin release and in the incidence of myocardial infarction) will translate into a better tissue perfusion and faster recovery as documented by reduced intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* written informed consent
* scheduled procedures

Exclusion Criteria:

* ongoing acute myocardial infarction
* cardiac troponin >1 ng/ml
* previous unusual response to an anesthetic
* use of sulfonylurea, theophylline or allopurinol
* thoracotomy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Composite endpoint or number of dead patients and/or number of patients requiring prolonged intensive care unit stay

SECONDARY OUTCOMES:
cardiac troponin release
incidence of perioperative myocardial infarction
time on mechanical ventilation
postoperative hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: giovanni landoni, MD, Principal Investigator — Vita-Salute University of Milano. Italy; elena bignami, MD, Study Director — Vita-Salute University of Milano, Italy
Locations (5):
- Italy (5):
  - Vita-Salute University, Milan
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Ospedaliera di Perugia (H Santa Maria della Misericordia), Perugia
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Università La Sapienza, Policlinico Umberto I, Roma, Roma

REFERENCES:
- [Background] Landoni G, Biondi-Zoccai GG, Zangrillo A, Bignami E, D'Avolio S, Marchetti C, Calabro MG, Fochi O, Guarracino F, Tritapepe L, De Hert S, Torri G. Desflurane and sevoflurane in cardiac surgery: a meta-analysis of randomized clinical trials. J Cardiothorac Vasc Anesth. 2007 Aug;21(4):502-11. doi: 10.1053/j.jvca.2007.02.013. Epub 2007 May 7. PMID 17678775
- [Background] Landoni G, Fochi O, Tritapepe L, Guarracino F, Belloni I, Bignami E, Zangrillo A. Cardiac protection by volatile anesthetics. A review. Minerva Anestesiol. 2009 May;75(5):269-73. Epub 2008 Nov 6. PMID 18987572
- [Background] Landoni G, Zangrillo A, Fochi O, Maj G, Scandroglio AM, Morelli A, Tritapepe L, Montorfano M, Colombo A. Cardiac protection with volatile anesthetics in stenting procedures. J Cardiothorac Vasc Anesth. 2008 Aug;22(4):543-7. doi: 10.1053/j.jvca.2008.02.020. Epub 2008 May 14. PMID 18662628
- [Background] Landoni G, Fochi O, Zangrillo A. Cardioprotection by volatile anesthetics in noncardiac surgery? No, not yet at least. J Am Coll Cardiol. 2008 Apr 1;51(13):1321; author reply 1321-2. doi: 10.1016/j.jacc.2007.12.020. No abstract available. PMID 18371566
- [Background] Landoni G, Calabro MG, Marchetti C, Bignami E, Scandroglio AM, Dedola E, De Luca M, Tritapepe L, Crescenzi G, Zangrillo A. Desflurane versus propofol in patients undergoing mitral valve surgery. J Cardiothorac Vasc Anesth. 2007 Oct;21(5):672-7. doi: 10.1053/j.jvca.2006.11.017. Epub 2007 Feb 22. PMID 17905272
- [Background] Tritapepe L, Landoni G, Guarracino F, Pompei F, Crivellari M, Maselli D, De Luca M, Fochi O, D'Avolio S, Bignami E, Calabro MG, Zangrillo A. Cardiac protection by volatile anaesthetics: a multicentre randomized controlled study in patients undergoing coronary artery bypass grafting with cardiopulmonary bypass. Eur J Anaesthesiol. 2007 Apr;24(4):323-31. doi: 10.1017/S0265021506001931. Epub 2006 Dec 8. PMID 17156509
- [Background] Guarracino F, Landoni G, Tritapepe L, Pompei F, Leoni A, Aletti G, Scandroglio AM, Maselli D, De Luca M, Marchetti C, Crescenzi G, Zangrillo A. Myocardial damage prevented by volatile anesthetics: a multicenter randomized controlled study. J Cardiothorac Vasc Anesth. 2006 Aug;20(4):477-83. doi: 10.1053/j.jvca.2006.05.012. PMID 16884976
- [Background] Landoni G, Zambon M, Zangrillo A. Reducing perioperative myocardial infarction with anesthetic drugs and techniques. Curr Drug Targets. 2009 Sep;10(9):858-62. doi: 10.2174/138945009789108837. Epub 2009 Sep 1. PMID 19538174
- [Background] Bignami E, Biondi-Zoccai G, Landoni G, Fochi O, Testa V, Sheiban I, Giunta F, Zangrillo A. Volatile anesthetics reduce mortality in cardiac surgery. J Cardiothorac Vasc Anesth. 2009 Oct;23(5):594-9. doi: 10.1053/j.jvca.2009.01.022. Epub 2009 Mar 19. PMID 19303327
- [Derived] Landoni G, Guarracino F, Cariello C, Franco A, Baldassarri R, Borghi G, Covello RD, Gerli C, Crivellari M, Zangrillo A. Volatile compared with total intravenous anaesthesia in patients undergoing high-risk cardiac surgery: a randomized multicentre study. Br J Anaesth. 2014 Dec;113(6):955-63. doi: 10.1093/bja/aeu290. Epub 2014 Sep 3. PMID 25186820
- See also: ITACTA (Italian Association of Cardiothoracic Anesthesiologists) — http://www.itacta.org